CLINICAL TRIAL: NCT06492096
Title: Relation Between Bibloc Mandibular Advancement Oral Appliance Used In Treatment of Obstructive Sleep Apnea and Tempromandibular Joint Health
Brief Title: Bibloc Mandibular Advancement Oral Device and Its Effect on TMJ Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M06050422
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMD Group (Active Comparator)
  Interventions: Device: Bibloc Mandibular Advancement device
- Non_TMD Group (Active Comparator)
  Interventions: Device: Bibloc Mandibular Advancement device

INTERVENTIONS:
Device: Bibloc Mandibular Advancement device — Each patient received a CAD/CAM designed Bibloc Mandibular Advancement device

SUMMARY:
The goal of this clinical trial is to learn if Mandibular Advancement Device( MAD) works to treat Obstructive sleep apnea in adults. It will also learn about the effect of the device on the Tempromandibular Joint Health . The main questions it aims to answer are:

Does MAD lower the number of apnoea and hypopnea participants suffer from during sleep? Would it cause any effect on TMJ health? Researchers will compare between a group of TMD patients with OSA to a non_TMD group of patients also with sleep apnea and both groups will receive a Bibloc MADplacebo (a look-alike substance that contains no drug) to see if it affect the TMJ health.

Participants will:

Wear MAD during sleep (at least 6 hours) every day for 6 months Visit the clinic once after the first week for checkups and adjustment of MAD If needed and then after 3 months and 6 months.

Polysomnography, MRI, and tmd screening was done before the appliance insertion and after 6 months of its insertion.

ELIGIBILITY:
Inclusion Criteria:

- Patients having obstructive sleep apnea syndrome (OSAS) as determined by polysomnography with mild to moderate apnea/hypopnea index ranging from 5 to 30 events per hour of sleep. ( As 5-15 events per hour is considered mild condition, 16-30 is considered moderate).(1)

2- Adequate nasal air flow capacity as determined by qualified otolaryngologist.

Exclusion Criteria:

* patients having Central sleep apnea events as determined by the polysomnography.

  2- patients having cardiovascular disease. 3- History of alcohol, narcotic or psychoactive medications. 4- Serious nasal passage obstructions or allergies. 5- Previous history of treatment with any type of obstructive sleep apnea oral appliances.

  6- Obese patients with BMI more than 30. 7- Missing more than five teeth (excluding third molar). 8- Allergy to acrylic resin.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Apnea/Hypopnea index | 6 months
  Number of apnea and hypopnea per hour of sleep

SECONDARY OUTCOMES:
Condylar disc position | 6 months
  It appears in MRI and measured before and after the appliance insertion
Joint space of TMJ | 6 months
  measurement of joint space was done for each patient on their MRI before and after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Mansoura university, Al Manşūrah, Ad Dakahlia, Egypt